CLINICAL TRIAL: NCT05284513
Title: Collaborative Approach to Reach Everyone With Familial Hypercholesterolemia (CARE-FH)
Acronym: CARE-FH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samuel Gidding, Professor, Geisinger Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021-0927; 1R61HL161775 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2022-03-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1 (Other): Phased rollout to clinic sites across the the Geisinger system using stepped wedge design
  Interventions: Behavioral: FH diagnosis program; Behavioral: Implementation strategy package: Develop and implement tools for quality monitoring; Behavioral: Implementation strategy package: Develop educational materials; Behavioral: Implementation strategy package: Conduct educational outreach visits; Behavioral: Implementation strategy package: Intervene with clinicians and patients to enhance; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) Implementation strategy package: Identify and prepare champions Clinical lipid champions; Behavioral: Implementation strategy package: Audit and provide feedback; Behavioral: Implementation strategy package: Stage implementation scale up
- Phase 2 (Other): Phased rollout to clinic sites across the the Geisinger system using stepped wedge design
  Interventions: Behavioral: FH diagnosis program; Behavioral: Implementation strategy package: Develop and implement tools for quality monitoring; Behavioral: Implementation strategy package: Develop educational materials; Behavioral: Implementation strategy package: Conduct educational outreach visits; Behavioral: Implementation strategy package: Intervene with clinicians and patients to enhance; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) Implementation strategy package: Identify and prepare champions Clinical lipid champions; Behavioral: Implementation strategy package: Audit and provide feedback; Behavioral: Implementation strategy package: Stage implementation scale up
- Phase 3 (Other): Phased rollout to clinic sites across the the Geisinger system using stepped wedge design
  Interventions: Behavioral: FH diagnosis program; Behavioral: Implementation strategy package: Develop and implement tools for quality monitoring; Behavioral: Implementation strategy package: Develop educational materials; Behavioral: Implementation strategy package: Conduct educational outreach visits; Behavioral: Implementation strategy package: Intervene with clinicians and patients to enhance; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) Implementation strategy package: Identify and prepare champions Clinical lipid champions; Behavioral: Implementation strategy package: Audit and provide feedback; Behavioral: Implementation strategy package: Stage implementation scale up
- Phase 4 (Other): Phased rollout to clinic sites across the the Geisinger system using stepped wedge design
  Interventions: Behavioral: FH diagnosis program; Behavioral: Implementation strategy package: Develop and implement tools for quality monitoring; Behavioral: Implementation strategy package: Develop educational materials; Behavioral: Implementation strategy package: Conduct educational outreach visits; Behavioral: Implementation strategy package: Intervene with clinicians and patients to enhance; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) Implementation strategy package: Identify and prepare champions Clinical lipid champions; Behavioral: Implementation strategy package: Audit and provide feedback; Behavioral: Implementation strategy package: Stage implementation scale up
- Phase 5 (Other): Phased rollout to clinic sites across the the Geisinger system using stepped wedge design
  Interventions: Behavioral: FH diagnosis program; Behavioral: Implementation strategy package: Develop and implement tools for quality monitoring; Behavioral: Implementation strategy package: Develop educational materials; Behavioral: Implementation strategy package: Conduct educational outreach visits; Behavioral: Implementation strategy package: Intervene with clinicians and patients to enhance; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) Implementation strategy package: Identify and prepare champions Clinical lipid champions; Behavioral: Implementation strategy package: Audit and provide feedback; Behavioral: Implementation strategy package: Stage implementation scale up

INTERVENTIONS:
Behavioral: FH diagnosis program — Uptake of screening, diagnosis, and initiation of care management for FH
Behavioral: Implementation strategy package: Develop and implement tools for quality monitoring — EHR tools to order labs, record results, and document FH care
Behavioral: Implementation strategy package: Develop educational materials — Education regarding guidelines for identification and treatment of FH
Behavioral: Implementation strategy package: Conduct educational outreach visits — Continuing medical education (CME) material for FH that is presented to
Behavioral: Implementation strategy package: Intervene with clinicians and patients to enhance — Notify patients simultaneously with clinicians about the need for screening
Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) Implementation strategy package: Identify and prepare champions Clinical lipid champions — Clinical lipid champions
Behavioral: Implementation strategy package: Audit and provide feedback — Provide aggregate level feedback to clinics on diagnosing FH
Behavioral: Implementation strategy package: Stage implementation scale up — Develop the timeline for the stepped-wedge rollout to primary care

SUMMARY:
Diagnosis rates of familial hypercholesterolemia (FH) are low in the United States, despite multiple guidelines and recommendations for screening and treatment of high cholesterol, to prevent heart attacks in those affected. Using a stepped-wedge design, the investigators plan to utilize tools from implementation science to improve uptake, acceptability, and sustainability of FH diagnostic programs in primary care settings. If successful, this study will provide tools generalizable to other health care systems to improve FH diagnosis rates.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is a common genetic disorder (prevalence 1 in 250) that requires lifelong sustained medical care. Evidence-based guidelines for screening and treatment for FH exist. These include universal screening of children ages 9-11, of adolescents ages 18-20, and of adults ages 40 and above; approved diagnostic tools including lipid panels and genetic testing; and recommendations for initiation of lipid lowering medication. FH diagnosis is currently made too late in life, often after a premature heart attack has occurred creating a care gap that results in excess cardiovascular morbidity and mortality. Diagnosing FH in the primary care setting would optimize treatment for individuals with FH and close this care gap. Utilizing tools from implementation science and human centered design, and by considering uptake, acceptability, and sustainability of programs related to FH care should improve earlier diagnosis. Implementation strategies that include insights from patients, clinicians, and healthcare systems are necessary. The long-term goal is to create an effective FH diagnosis program that is practical and sustainable in the real-world setting. The main objective of this project is to determine the uptake of an FH diagnosis program integrated into primary care practices to promote early identification of adult and pediatric patients that is generalizable to other healthcare settings. The research question is, does using a multi-level implementation strategy package, designed to address the specific needs of patients, clinicians, and healthcare systems, improve the diagnosis and activation of care management for individuals with FH. The specific aims are to: 1) to design a clinical trial to assess multi-level implementation strategies for improving FH diagnosis in an integrated health system, 2) compare FH diagnosis rates among primary care clinicians who receive the implementation strategy package versus those who do not, 3) to measure implementation success of an organized FH diagnosis program, and 4) to explore patient-related service and health outcomes related to an FH diagnosis program.

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinicians (pediatrician, community medicine, internal medicine) in the Geisinger Healthcare System

Exclusion Criteria:

* None

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
FH diagnosis rate (Aim 2) | Up to 45 months
  FH diagnosis rate, is achieving both the scheduling of a clinic visit and evidence the clinician, at that visit, has completed evidence-based FH diagnostic evaluation, defined as completing one of: using the FH clinic note to document care, adding FH diagnosis on the problem list, using the FH smart-set (or ordered a genetic test for FH), making a referral to the lipid clinic, or starting a statin for an evidence-based indication
Acceptability (Aim 3) | Month 9, 12, 18, 24, 30, 36, 42
  Clinician and patient satisfaction and self-efficacy with the FH diagnosis program
Timeliness (Aim 4) | Up to 45 months
  Time to FH screen, time to diagnostic evaluation, time to statin initiation

SECONDARY OUTCOMES:
Initiation medication use (Aim 2) | Up to 45 months
  Initiation of lipid lowering medication by healthcare clinician
Lipid measurement (Aim 2) | Up to 45 months
  Order of a lipid panel
Genetic testing (Aim 2) | Month 9, 12, 18, 24, 30, 36, 42
  Order of a genetic test for FH
Problem list diagnosis of FH (Aim 2) | Up to 45 months
  Clinician adds diagnosis of FH to the patients problem list in the electronic health record
FH smartset (Aim 2) | Month 9, 12, 18, 24, 30, 36, 42
  Clinician uses and completes all field of the FH smartset
Best Practice Alert (Aim 2) | Up to 45 months
  Clinician adheres to and acts on recommendation in the Best Practice Alert
FH Clinic Note (Aim 2) | Up to 45 months
  Clinician completes the FH clinic note
Fidelity (Aim 3) | Up to 45 months
  Documentation of adaptations to the FH diagnosis program
Cost (Aim 3) | Up to 45 months
  Cost to implement the implementation strategy package
Function (Aim 4) | Up to 45 months
  Return of genetic result to patient (if ordered and patient undergoes testing)
Function (Aim 4) | Up to 45 months
  Reduction in lipid level from baseline to end of the study period
Function (Aim 4) | Up to 45 months
  Patient side effects to medications

CONTACTS AND LOCATIONS:
Overall Officials: Laney K Jones, PharmD, MPH, Principal Investigator — Geisinger Clinic; Samuel S Gidding, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Multiple Locations, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Available upon request from PIs

REFERENCES:
- [Derived] Jones LK, Romagnoli KM, Schubert TJ, Clegg K, Kirchner HL, Hu Y, Cawley D, Norelli V, Williams MS, Gidding SS, Rahm AK. Using implementation science to develop a familial hypercholesterolemia screening program in primary care: The CARE-FH study. J Clin Lipidol. 2024 Mar-Apr;18(2):e176-e188. doi: 10.1016/j.jacl.2024.01.001. Epub 2024 Jan 4. PMID 38228467